CLINICAL TRIAL: NCT03957499
Title: Analgesic Efficacy of Fascia Iliaca Compartment Block With Bupivacaine Versus Bupivacaine With Dexamethasone or Magnesium Sulphate for Dynamic Hip Screw Surgeries Randomized Double Blinded Comparative Study
Brief Title: Analgesic Efficacy of Fascia Iliaca Compartment Block
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samaa Rashwan (Other)
Responsible Party: Sponsor-Investigator, Samaa Rashwan, Principal Investigator, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Beni-Suef Faculty of Medicine
Record Dates: First submitted 2019-05-13; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine; Dexamethasone; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The anesthetists who will prepare the drug and who will collect the data will be blinded to the study protocol
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the control group (Placebo Comparator): Ultrasound guided fascia iliaca compartment block (FICB) will be performed using 28 ml bupivacaine 0.25% + 2 ml of normal saline (total volume 30 ml).(
  Interventions: Drug: Bupivacaine
- Group dexamethasone/Bupivacaine: (Active Comparator): Ultrasound guided fascia iliaca compartment block (FICB) will be performed using with 28 ml bupivacaine 0.25% + 2 ml dexamethasone (8mg) (total volume 30 ml).(
  Interventions: Drug: Dexamethasone/bupivacaine
- Group Magnesium sulphate/Bupivacaine (Active Comparator): Ultrasound guided fascia iliaca compartment block (FICB) will be performed using 28 ml bupivacaine 0.25% + 2 ml magnesium sulphate (200mg) (total volume 30 ml).
  Interventions: Drug: Magnesium Sulfate/bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Ultrasound guided fascia iliaca compartment block (FICB) will be performed using 28 ml bupivacaine 0.25% + 2 ml of normal saline (total volume 30 ml).(
  Other Names: Marcain
  Arms: the control group
Drug: Dexamethasone/bupivacaine — Ultrasound guided fascia iliaca compartment block (FICB) will be performed with 28 ml bupivacaine 0.25% + 2 ml dexamethasone (8mg) (total volume 30 ml)d using
  Arms: Group dexamethasone/Bupivacaine:
Drug: Magnesium Sulfate/bupivacaine — Ultrasound guided fascia iliaca compartment block (FICB) will be performed using 28 ml bupivacaine 0.25% + 2 ml magnesium sulphate (200mg) (total volume 30 ml).
  Arms: Group Magnesium sulphate/Bupivacaine

SUMMARY:
The aim of this study is to evaluate the analgesic efficacy of fascia iliaca compartment block using bupivacaine versus bupivacaine with dexamethasone or magnesium sulphate for dynamic hip screw surgery under spinal anesthesia.

The primary outcome will be the duration of effective analgesia from FICB till the first analgesic dose is required,the secondary outcomes will be the severity of postoperative pain as will be assessed by the visual analogue scale and the total dose of pethidin for rescue analgesia.

DETAILED DESCRIPTION:
Different modes of analgesia are given prior to neuraxial blockade for pain relief like non-steroidal anti-inflammatory drugs (NSAID), opioids and peripheral nerve blocks such as, femoral nerve block, 3 in 1 block or fascia iliaca compartment block (FICB).

FICB is believed to be most beneficial compared to other procedures because of its safety and efficacy . FICB provides blockage of at least two of the three major nerves that supply the medial, anterior and lateral thigh with one simple injection, namely the femoral and lateral femoral cutaneous nerves.

FICB is an anterior approach to the lumbar plexus. The pop technique using fascial click had a low success rate of 35% - 47% .However, as the FICB was performed under real-time ultrasound guidance, the success rate was increased up to 82- 87%, leading to an increased interest in FICB as a postoperative analgesia option for hip and knee surgical procedures .

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology physical status (ASA) I & II of both sex.
* Age between 20 and 70 years.
* Patients with traumatic hip fracture presenting for elective or emergency dynamic hip screw (DHS) fixation under spinal anesthesia.

Exclusion Criteria:

* Patient refused to give consent
* Patients with history of allergy to dexamethasone, magnesium sulphate or bupivacaine.
* Patients with contraindications to spinal anesthesia.
* Previous surgery in the affected hip, infection at the injection site, multiple fractures.
* Peripheral neuropathy.
* Use of analgesics within 8 hours before the spinal block.
* Inguinal hernia, and femoral artery graft.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Analgesia | duration from the end of surgery till the first time to ask for post operative analgesia within the first 12 hours after surgery
  the duration of effective analgesia will be considered as the duration after performing the FICB till the patient ask for first analgesic dose ,in this case pethidin 25 mg will be given intravenously

CONTACTS AND LOCATIONS:
Overall Officials: Samaa Rashwan, MD, Principal Investigator — Assisstant proffesor of anesthesia
Locations (1):
- Beni-Suef University Hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No